CLINICAL TRIAL: NCT02867358
Title: A Multi-center, Randomized, Double-blind, and Placebo-controlled Phase II Clinical Study to Investigate the Safety and Efficacy of Two Doses of KT07 Compared to Placebo in Subjects With Acute Uncomplicated Influenza
Brief Title: A Clinical Trial of KT07 Capsule in the U.S.A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yiling Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KT07-US-01
Record Dates: First submitted 2016-08-10; First posted 2016-08-15 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Influenza, Human
Keywords: acute uncomplicated influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High dose of KT07 capsule (Active Comparator): It will assess about 140 subjects with influenza at high dose KT07 (6 capsules each time, bid).
  Interventions: Drug: KT07 Capsule
- Low dose of KT07 capsule (Active Comparator): It will assess about 140 subjects with influenza at low dose KT07 (4 capsules of KT07 + 2 capsules of placebo each time, bid).
  Interventions: Drug: KT07 Capsule; Other: Placebo
- Placebo (Placebo Comparator): It will assess 140 subjects with influenza using 6 capsules of placebo each time, bid as control.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KT07 Capsule
  Other Names: Lianhua Qingwen Capsule
  Arms: High dose of KT07 capsule; Low dose of KT07 capsule
Other: Placebo
  Arms: Low dose of KT07 capsule; Placebo

SUMMARY:
The purpose of this study is to investigate clinical efficacy of KT07 capsule in alleviation of fever and other symptoms including nasal congestion, sore throat, cough, aches and pains, fatigue, headache, chills or sweats in subjects with acute uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria

1. Subjects with acute uncomplicated influenza with oral temperature ≥ 37.8 ℃ (100.04 °F); plus at least one respiratory symptom (nasal congestion, sore throat, cough); and at least one constitutional symptom (aches or pains, fatigue, headache, chills or sweats). If antipyretics were taken, may wait at least 4 hours after dosing to determine if a qualifying temperature is observed.
2. Subjects with RIDT confirmed influenza infection.
3. Onset of symptoms less than 48 hours before Visit 1 (Screening; study drug administration visit). The onset of symptoms is defined as either:

   * Time of the first increase in body temperature to ≥ 37.8 ℃ (100.04 °F); or
   * Time when the subject experiences at least one general or respiratory symptom.
4. Age 18 to 65 years old.
5. Subjects who are able to understand and willing to sign the informed consent form (ICF).
6. All female subjects of child-bearing potential must have a negative urine pregnancy test result. All female subjects of child-bearing potential and male subjects and their spouse/partner must agree to use a medically acceptable method of contraception (e.g., abstinence, an intrauterine device, a double barrier method such as condom + spermicide or condom + diaphragm with spermicide, a contraceptive implant, an oral contraceptive or have a vasectomized partner with confirmed azoospermia) throughout the entire study period, and for 30 days for females and 90 days for males after study drug discontinuation.

Exclusion Criteria

1. Subjects with severe influenza virus infection requiring inpatient treatment.
2. Subjects with concurrent infections requiring systemic antimicrobial and/or antiviral therapy at the time of screening.
3. Subjects who have any of the following documented conditions: uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg), diabetes, asthma (any current or recent, not childhood if resolved), COPD (any), cardiac, hepatic, renal (including eGFR<60) and hematopoietic disorders, bleeding tendency or hemorrhagic disease, neurological system disease, compromised immune system (including patients receiving immunosuppressant therapy, or those with cancer within the past 5 years or human immunodeficiency virus [HIV] infection), endocrine disorders (including thyroid disorders).
4. Subjects with anatomical nasal obstruction or gross anatomical abnormalities. For example, nasal polyps or significant nasal septal deviation.
5. Clinically obese subjects with BMI≥40.
6. Subjects with recent history (within 1 year) of alcoholism or substance abuse.
7. Received influenza vaccine within 21 days.
8. Participation in other clinical trial within 1 month, or during the study.
9. Pregnant or breast-feeding female subjects
10. Allergy or known allergy to components of study medication.
11. Subjects who took a monoamine oxidase inhibitor (MAOI) within 2 weeks prior to enrollment.
12. Previous history of difficulty swallowing capsules.
13. Any other associated disease or condition which, in the opinion of the investigator, might restrict or impede participation in the study or affect the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
To investigate the improvement in reducing the duration of illness compared to placebo. | Up to 19 days
  Duration of illness is defined as: the length of time to alleviation of all symptoms.
  The duration of alleviation is calculated from time 0 (first administration of study medication) to the time at which symptom is alleviated.

SECONDARY OUTCOMES:
The reduction in duration of alleviation of individual symptom | Up to 19 days
  From time zero to the time at which the symptom is less than or equal to mild and stable for at least 24 hours
Quality of life assessment | Up to 19 days
  Based on the self-assessment questionnaire

OTHER OUTCOMES:
Influenza viral shedding from baseline to Day 3 and Day 6 post treatment initiation during KT07 treatment | Day 1 & 3 & 6
  Reduction in viral shedding; Influenza viral AUC

CONTACTS AND LOCATIONS:
Overall Officials: Xuedong Gao, MD, Study Director — Yiling Pharmaceutical Inc.
Locations (81):
- United States (81):
  - Central Alabama Research, Birmingham, Alabama
  - Parkway Medical Center, LLC, Birmingham, Alabama
  - Cahaba Research, Inc., Birmingham, Alabama
  - David Wever, Pelham, Alabama
  - Alliane Urgent Care, Tolleson, Arizona
  - Orange County Research Institute, Anaheim, California
  - Hope Clinical Research, Inc., Canoga Park, California
  - Core Health Care Group, Cerritos, California
  - Aviva Research, Escondido, California
  - Lalla-Reddy Medical Corp., Fountain Valley, California
  - Research Center of Fresno, Inc., Fresno, California
  - Ark Clinical Research, Long Beach, California
  - Long Beach Clinical Trials Services, Inc, Long Beach, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - IMD Medical Group, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - MD Strategies Research Centers, San Diego, California
  - Empire Clinical Research, Upland, California
  - Cherry Creek Family Practice, PLLC, Denver, Colorado
  - Urgent Care-Denver, Denver, Colorado
  - Clinical Research Consulting, Milford, Connecticut
  - Comprehensive Psychiatric Center, Norwich, Connecticut
  - Doral Medical Research, Doral, Florida
  - Finlay Medical Research Corp., Miami, Florida
  - Panamerican Health Center, Inc., Miami, Florida
  - AppleMed Reseach, Inc., Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Sweet Hope Research Specialty, Inc, Miami Lakes, Florida
  - Sunrise Medical Research, Tamarac, Florida
  - Sunrise Medical Research, West Palm Beach, Florida
  - Southeast Clinical Research, Williston, Florida
  - Invocare (Savannah GA location), Rincon, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - The Blackfoot Medical Center - Blackfoot, Blackfoot, Idaho
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - Horizon Research Group of Opelousas, LLC, Eunice, Louisiana
  - Centex Studies, Inc, Lake Charles, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Romedica LLC, Rochester, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Red Rock Clinical Research, LLC, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - New York Clinical Trials, Manhattan, New York
  - Carolina Research Center, Inc, Shelby, North Carolina
  - Ardmore Family Practice, Winston-Salem, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - META Medical Research Institute, LLC, Dayton, Ohio
  - Medical Research International, Oklahoma City, Oklahoma
  - Detweiler Family Medicine, Lansdale, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - American Family Care Urgent Care, Chattanooga, Tennessee
  - Clinical Research Solutions, LLC, Franklin, Tennessee
  - Clinical Research Solutions, LLC, Jackson, Tennessee
  - Clinical Research Solutions, LLC, Nashville, Tennessee
  - Clinical Research Solutions, LLC, Smyrna, Tennessee
  - Clinical Research Solutions, LLC, Spring Hill, Tennessee
  - Premier Family Physicians, Austin, Texas
  - Pioneer Research Solutions, Beaumont, Texas
  - Family Medicine Associates of Texas, Carrollton, Texas
  - Corpus Christi Family Wellness, Corpus Christi, Texas
  - Northwest Med Care, Cypress, Texas
  - City Doc Urgent Care, Dallas, Texas
  - Centex Studies, Inc., Houston, Texas
  - Centex Studies, Inc., McAllen, Texas
  - Village Health Partners, Plano, Texas
  - Quaity Assurance Research Center, San Antonio, Texas
  - Bandera Family Health Clinic, San Antonio, Texas
  - Wade Family Medicine, Bountiful, Utah
  - J. Lewis Research, Inc./ Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc./ FirstMed East, Salt Lake City, Utah
  - CopperView Medical Center, South Jordan, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Clinical Research Partners, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No